CLINICAL TRIAL: NCT00901433
Title: Self Operating of the Personal WheezoMeter by Intended Users - A Usability Study
Status: Completed | Type: Observational
Sponsor: KarmelSonix Ltd. (Industry)
Responsible Party: Dr. Hanna Levy - Director of clinical studies, KarmelSonix Ltd
Other Study IDs: KSI-PW-US-01
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Last update posted 2009-06-24 (Estimated); Status verified 2009-05

CONDITIONS: Asthma
Keywords: Asthma; Wheeze Rate; Respiratory Function Tests
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Usability study of the Personal Wheezometer
  Interventions: Device: Personal WheezoMeter

INTERVENTIONS:
Device: Personal WheezoMeter — pulmonary sounds analyzer

SUMMARY:
The NAEPP (National Asthma Education and Prevention Program) guidelines recommend that spirometry be performed on patients with asthma because they serve as an objective measure of airway obstruction. Unfortunately, most children under 5 years of age are unable to perform a forced expiratory maneuver making conventional spirometry unavailable in this age group in most venues. Furthermore, other population groups such as retarded people, elderly or physically handicapped share the same difficulty.

Karmel Sonix Ltd has developed the Personal WheezoMeter a hand-held pulmonary sounds analyzer that utilizes contact sensors to acquire, amplify, filter, record and quantify the presence of wheezing. This usability study was designed to test independent home use and device interface effectiveness of the Personal WheezoMeter in order to validate its safe and effective use by intended users.

ELIGIBILITY:
Inclusion Criteria:

* Male/female age 18 years and up.
* Subject is diagnosed as an asthmatic, or subject is parent/guardian of an asthmatic child age under 18 years.
* Subject understands the study procedure.
* Subject is able to read the User Manual.
* Signed Informed Consent form
* Compliance with study requirements.

Exclusion Criteria:

* Major physical, motor, mental, behavioral, or psychiatric limitations.
* Concurrent additional major illness.
* Subject objects to the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male/Female participants ages 18 and up that were either diagnosed as an asthmatic or are parent/guardian of an asthmatic child age under 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Safety will be evaluated by success rate of task performance. | At the end of the study meeting

SECONDARY OUTCOMES:
Number of questions addressed to the investigator required by the participant in order to complete tasks. | during the study
User satisfaction will be evaluated by questionnaire that focuses on subjective impressions regarding usability and potential safety problems. | At the end of the study meeting.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Levy, Dr., Study Director — KarmelSonix Ltd.
Locations (1):
- RAMBAM Health Care Campus, Haifa, Israel